CLINICAL TRIAL: NCT01612598
Title: Feasibility of a Palliative Care Intervention for Patients on Phase 1 Clinical Trials
Brief Title: Palliative Care Intervention in Patients With Solid Tumors Participating in Phase I Clinical Trials
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 12123; NCI-2012-00887 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2012-06-04; First posted 2012-06-06 (Estimated); Last update posted 2014-01-31 (Estimated); Status verified 2014-01

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
MeSH Terms: interventions — Counseling; Early Intervention, Educational; Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Supportive Care (PCI) (Experimental): PCI PART I: Patients undergo comprehensive PC assessment based on baseline data and complete goals of care discussion.
  PCI PART II: Following the first dose of phase I investigational treatment, patients meet with the IDT, where PC recommendations are made. This is followed by two patient educational sessions that will cover QOL-related domains, including physical, social, emotional, and spiritual well-being. Supportive care referrals are made based on IDT recommendations.
  Interventions: Other: counseling intervention; Procedure: quality-of-life assessment; Other: questionnaire administration; Other: educational intervention

INTERVENTIONS:
Other: counseling intervention — Undergo PCI
  Other Names: counseling and communications studies
Procedure: quality-of-life assessment — Ancillary studies
  Other Names: quality of life assessment
Other: questionnaire administration — Ancillary studies
Other: educational intervention — Undergo PCI
  Other Names: intervention, educational

SUMMARY:
Patients enrolled in phase I clinical trials could potentially benefit from palliative care concurrently, yet limited evidence is available to support such a change in care. The primary purpose of this study is to test the feasibility of a palliative care intervention (PCI) for patients participating in a phase I therapeutic clinical trial

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Describe the feasibility of implementing a PCI for patients on phase I clinical trials (study accrual and retention).

II. Describe the initial impact of a PCI on key patient outcome measures (quality of life [QOL], psychological distress, satisfaction with communication, symptom intensity, symptom distress, and patient satisfaction) over time.

OUTLINE:

PCI PART I: Patients undergo comprehensive palliative care (PC) assessment based on baseline data and complete goals of care discussion.

PCI PART II: Following the first dose of phase I investigational treatment, patients meet with the interdisciplinary team (IDT), where PC recommendations are made. This is followed by two patient educational sessions that will cover QOL-related domains, including physical, social, emotional, and spiritual well-being. Supportive care referrals are made based on IDT recommendations.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with solid tumors who are being assessed for participation in phase I clinical trials of investigational cancer therapies
* Able to read or understand English
* Ability to read and/or understand the study protocol requirements, and provide written informed consent

Exclusion Criteria:

* Patient diagnosed with hematologic or brain cancers

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2012-07; Primary Completion 2013-06 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Study accrual and retention | 8 weeks
Change in psychological distress assessed using Distress Thermometer | Baseline to 8 weeks
  One-way repeated measure of Analysis of Covariance (ANCOVA), controlling for baseline scores and testing for within subjects change over time (4 weeks and 8 weeks) will be conducted to examine the PCI's impact on each of the outcome measures.
Change in satisfaction with communication assessed using Satisfaction with Communication Tool | Baseline to 8 weeks
  One-way repeated measure of ANCOVA, controlling for baseline scores and testing for within subjects change over time (4 weeks and 8 weeks) will be conducted to examine the PCI's impact on each of the outcome measures.
Change in QOL using Functional Assessment of Cancer Therapy- General (FACT-G) and Functional Assessment of Chronic Illness Therapy- Spirituality (FACT-Sp-12) | Baseline to 8 weeks
  Multivariate ANCOVAs (MANCOVAs) will be used at 4 and 8 weeks to examine the PCI's impact on QOL and symptom intensity and distress due to the multiple subscales in these two instruments.
Change in symptom intensity and distress using Memorial Symptom Assessment Scale (MSAS) | Baseline to 8 weeks
  MANCOVAs will be used at 4 and 8 weeks to examine the PCI's impact on QOL and symptom intensity and distress due to the multiple subscales in these two instruments.

CONTACTS AND LOCATIONS:
Overall Officials: Betty Ferrell, Principal Investigator — City of Hope Medical Center
Locations (2):
- United States (2):
  - City of Hope Medical Center, Duarte, California
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins Hospital, Baltimore, Maryland

REFERENCES:
- [Derived] Ferrell B, Chung V, Hughes MT, Koczywas M, Azad NS, Ruel NH, Knight L, Cooper RS, Smith TJ. A Palliative Care Intervention for Patients on Phase 1 Studies. J Palliat Med. 2021 Jun;24(6):846-856. doi: 10.1089/jpm.2020.0597. Epub 2020 Oct 27. PMID 33103938